CLINICAL TRIAL: NCT01465620
Title: Dietetic and Hygiene Measures in Metabolic Neuropathies: the Neurodiet Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Sophie Ng Wing Tin, Investigator, clinical doctor, Henri Mondor University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM01
Record Dates: First submitted 2011-10-31; First posted 2011-11-07 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Nervous System Diseases; Diabetic Polyneuropathy; Metabolic Syndrome X
Keywords: Peripheral Nervous System Diseases; Diabetic Polyneuropathy; Metabolic Syndrome X
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetic Neuropathies; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaching (Experimental): active hygienic-dietetic coaching
  Interventions: Behavioral: hygienic-dietetic measures
- control (Active Comparator): reference hygienic-dietetic recommendations
  Interventions: Behavioral: hygienic-dietetic measures

INTERVENTIONS:
Behavioral: hygienic-dietetic measures — Therapeutic education about hygienic-dietetic measures followed by a 5 minutes phone call per week during 3 months
  Arms: Coaching
Behavioral: hygienic-dietetic measures — Therapeutic education about hygienic-dietetic measures followed by only one phone call
  Arms: control

SUMMARY:
Metabolic disorders such as diabetes mellitus, glucose intolerance and possibly metabolic syndrome can induce a peripheral neuropathy. To investigate the effect of physical training and diet education on neuropathic symptoms and neurophysiological parameters of patients with metabolic neuropathies.

DETAILED DESCRIPTION:
Metabolic disorder such as diabetes mellitus, glucose intolerance and possibly metabolic syndrome can induce a peripheral neuropathy. The objectives of the present study are to investigate:

1. the effect of physical training and diet education on neuropathic symptoms and neurophysiological parameters
2. the best coaching modality of education.

This will be a prospective single blind study (blinded evaluator). Patients will be randomly assigned in two groups. The first group will have a one-day therapeutic education program followed by a 5-minutes phone call every week for 3 months. The second group will have the same one-day therapeutic education program that will be followed by an unique one-hour phone call. During the one-day therapeutic education program and the phone calls, hygienic rules (ie physical activities) and dietetic regimen advices will be given to patients. Evaluation will be done at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and neurophysiologic neuropathy (clinical signs of neuropathy and at least two low sensory nerve action potential (superficial peroneal and sural nerves))
* Metabolic disorder: Glucose disorder (diabetes mellitus or glucose intolerance) or metabolic syndrome
* Clinical signs for less than 2 years
* No therapeutic modification in the last 3 months
* Possibility to delay any drug modification during 3 months

Exclusion Criteria:

* Non metabolic neuropathy
* Serious diabetic complication
* Renal failure (creatinine clearance<60ml/min)
* Sensory neuronopathy
* Contra-indication to physical activity
* Type 1 diabetes mellitus
* No written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in NTSS6 score at 3 months | 3 months
  Change from Baseline in NTSS6 score at 3 months (Bastyr EJ, 3rd, Price KL, Bril V. Development and validity testing of the neuropathy total symptom score-6: questionnaire for the study of sensory symptoms of diabetic peripheral neuropathy. Clin Ther. 2005 Aug;27(8):1278-94)

SECONDARY OUTCOMES:
clinical global impression of change | 3 months
change from baseline of sensory nerve action potential and sensory and motor nerve velocity | 3 months
  change from baseline of sensory nerve action potential and sensory and motor nerve velocity at 3 months
change from baseline of thermal and vibration thresholds | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alain Créange, MD PhD, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Hôpital Henri Mondor, Créteil, France